CLINICAL TRIAL: NCT04863937
Title: Distal Thigh Compression Garment Improves Knee Control and Safety Perceptions During Single Leg Triple Hop for Distance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spalding University (Other)
Responsible Party: Principal Investigator, John Nyland, Professor, Spalding University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REC-0118-2
Record Dates: First submitted 2021-04-21; First posted 2021-04-28 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Neuromuscular Control
Keywords: Dynamic Knee Stability

STUDY DESIGN:
Intervention Model Description: This study measured knee frontal plane projection angle (FPPA) and sports safety and performance perceptions of female athletes during a single leg triple hop for distance for 3 conditions (standard knee sleeve, no device and distal thigh compression garment (DTCG)).
Masking Description: Devices were used in a randomized order. The outcomes assessor evaluated device differences based on device numerical assignment..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Randomized Comparison of Knee Sleeve, Distal Thigh Compression Garment and No Device (Experimental): Randomized Comparison of Knee Sleeve, Distal Thigh Compression Garment and No Device
  Interventions: Device: Distal Thigh Compression Garment, Knee Sleeve

INTERVENTIONS:
Device: Distal Thigh Compression Garment, Knee Sleeve — Randomized Comparison of Knee Sleeve, Distal Thigh Compression Garment and No Device

SUMMARY:
This study measured knee frontal plane projection angle (FPPA) and sports safety and performance perceptions of female athletes during a single leg triple hop for distance for 3 conditions (standard knee sleeve, no device and distal thigh compression garment (DTCG)). The hypothesis was that the DTCG group would display superior dynamic knee valgus FPPA compared to the standard knee sleeve and no device groups.

DETAILED DESCRIPTION:
Eighteen healthy college athletes participated in this prospective cohort study with a randomized device order. FPPA was measured during single leg triple hop for distance using two-dimensional biomechanical techniques to estimate dynamic knee valgus loading. A 10-cm visual analog scale survey collected data regarding subject perceived knee control, sports movement capability and overall satisfaction for each condition. Pearson correlations delineated knee valgus, safety and performance relationship perceptions (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* College athletes
* ≥ 18 years

Exclusion Criteria:

* Knee injury history
* Any current lower extremity injury

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female college athletes
Enrollment: 18 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Frontal Plane Knee Projection Angle | Immediately after the intervention
  Frontal plane tibio-femoral alignment at single leg triple hop completion
Subject Confidence in Sports Safety and Performance Perceptions | Immediately after the intervention
  10-cm Visual Analog Confidence Scale for Sports Movement Capability and Safety Perceptions. Minimum value = 0. Maximum value = 100. Higher score equals greater confidence.

CONTACTS AND LOCATIONS:
Overall Officials: John Nyland, Study Director — Spalding University
Locations (1):
- Kosair Charities College of Health and Natural Sciences, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Data collection has been completed. Information will be presented in published manuscript.